CLINICAL TRIAL: NCT00998738
Title: The Use of Calcium and Magnesium for Prevention of Ixabepilone Induced Peripheral Neuropathy: A Phase III Double-Blind Placebo Controlled Study
Brief Title: Calcium and Magnesium in Preventing Peripheral Neuropathy Caused by Ixabepilone in Patients With Breast Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of accrual
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RC08CC; NCI-2009-01229 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RC08CC (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Results first posted 2013-08-29 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2015-11

CONDITIONS: Neuropathy; Pain; Recurrent Breast Carcinoma; Stage IV Breast Cancer
MeSH Terms: conditions — Pain; Breast Neoplasms | interventions — Calcium Gluconate; Calcium; Magnesium Sulfate; ixabepilone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (calcium gluconate, magnesium sulfate) (Experimental): Patients receive calcium gluconate and magnesium sulfate IV over 30 minutes immediately before and after each ixabepilone administration.
  Interventions: Drug: Calcium Gluconate; Drug: Magnesium Sulfate; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Ixabepilone
- Arm II (placebo) (Placebo Comparator): Patients receive placebo IV over 30 minutes immediately before and after each ixabepilone administration.
  Interventions: Other: Placebo; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Ixabepilone

INTERVENTIONS:
Drug: Calcium Gluconate — Given IV
  Other Names: Calcium D-gluconate; Calglucon
  Arms: Arm I (calcium gluconate, magnesium sulfate)
Drug: Magnesium Sulfate — Given IV
  Other Names: Magnesium SO4; Magnesium Sulfate whiskers
  Arms: Arm I (calcium gluconate, magnesium sulfate)
Other: Placebo — Given IV
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Ixabepilone — Given IV
  Other Names: IXEMPRA

SUMMARY:
This randomized phase III trial studies calcium and magnesium to see how well they work in preventing peripheral neuropathy caused by ixabepilone in patients with breast cancer. Giving calcium together with magnesium may stop or delay the development of peripheral neuropathy in patients with cancer who are receiving treatment with ixabepilone. It is not yet known whether calcium and magnesium are effective in preventing peripheral neuropathy caused by ixabepilone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare ixabepilone-induced peripheral neuropathy (sensory) as measured by European Organization for Research and Treatment of Cancer (EORTC) Quality of life Questionnaire (QLQ)-Chemotherapy-Induced Peripheral Neuropathy (CIPN)20 sensory subscale between calcium (Ca) Magnesium (Mg) and placebo arms.

SECONDARY OBJECTIVES:

I. To compare the incidence of CTCAE measured grade 2+ and/or grade 3+ peripheral neuropathy between CaMg and placebo arms.

II. To compare the times to onset of CTCAE measured grade 2+ and/or grade 3+ peripheral neuropathy between CaMg and placebo arms.

III. To compare the proportion of patients requiring ixabepilone dose reductions and/or stopping ixabepilone secondary to peripheral neuropathy (sensory) between CaMg and placebo arms.

IV. To assess the toxicity of CaMg in this situation. V. To document the incidence and severity of the acute pain syndrome (APS, commonly known as arthralgias/myalgias) induced by ixabepilone.

VI. To evaluate whether CaMg will decrease the acute pain syndrome (APS). VII. To evaluate the incidence and characteristics of, and change in, ixabepilone-APS over several cycles.

VIII. To evaluate the association between the ixabepilone-APS and eventual chemotherapy-induced neuropathy.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive calcium gluconate and magnesium sulfate IV over 30 minutes immediately before and after each ixabepilone administration.

ARM II: Patients receive placebo IV over 30 minutes immediately before and after each ixabepilone administration.

After completion of study treatment, patients are followed up monthly for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo cancer treatment for metastatic breast cancer (weekly or once every three weeks) with ixabepilone with no prior exposure to ixabepilone and no more than 2 prior chemotherapy regimens for metastatic disease
* Serum calcium =< 1.2 x upper normal limit (UNL)
* Serum magnesium =< UNL
* Serum creatinine =< 1.5 x UNL
* Ability to sign informed consent and understand the nature of a placebo-controlled trial
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0, 1, or 2
* Ability to complete questionnaire(s) by themselves or with assistance
* Life expectancy >= 4 months
* Presence of a central line

Exclusion Criteria:

* Pre-existing history of peripheral neuropathy >= grade 2 (National Cancer Institute [NCI] CTCAE Active Version) due to any cause (chemotherapy, diabetes, alcohol, toxin, hereditary, etc.)
* Concurrent treatment with anticonvulsants, tricyclic antidepressants, or other neuropathic pain medications agents such as carbamazepine, phenytoin, valproic acid, gabapentin, lamotrigine, topical lidocaine patch, capsaicin cream, etc., or any other treatments specifically for prevention or treatment of neuropathy
* Other medical conditions, which in the opinion of the treating physician/allied health professional would make this protocol unreasonably hazardous for the patient
* Any of the following:

  * Pregnant women
  * Nursing women
  * Women of childbearing potential (per physician judgment)
* Diagnosed diabetes requiring insulin or oral hypoglycemic medications
* Receiving digoxin or digitoxin
* History of heart block (any degree)
* Current treatment for arrhythmias
* Concurrent treatment with other neuropathic chemotherapy agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-11; Primary Completion 2010-07 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Loprinzi, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One participant was recruited between November 2009 and July 2010 at Mayo Clinic. This trial was terminated in July 2010 due to lack of accrual. Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Period: Overall Study
Arm/Group | Overall
Started | 1
Completed | 0
Not Completed | 1
Not completed — Uknown | 1

BASELINE CHARACTERISTICS:
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Overall
Number analyzed (Participants) | 0
Age, Categorical [Count of Participants; unit: Participants]
Age, Continuous [Mean (Standard Deviation); unit: years]
Sex: Female, Male [Count of Participants; unit: Participants]
Region of Enrollment [Number; unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Chemotherapy-induced Peripheral Neuropathy Between Calcium With Magnesium (CaMg) and Placebo Arms, as Measured by the Sensory Subscale of EORTC QLQ-CIPN20
Description: European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Chemotherapy-Induced Peripheral Neuropathy Module (EORTC QLQ-CIPN20) sensor subscale score was calculated following the standard scoring algorithm and was transformed to a 0 to 100 scale with 0=Low QOL and 100=Best QOL for data analysis.
Time Frame: During the first 18 weeks of ixabepilone-based therapy
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Overall
Number analyzed (Participants) | 0

2. Secondary Outcome: Percentage of Patients With Grade 2+ and/or Grade 3+ Neurotoxicity as Measured by NCI CTCAE Active Version Neuropathy Scale
Time Frame: Up to 12 months from initiation of ixabepilone
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Overall
Number analyzed (Participants) | 0

3. Secondary Outcome: Time to Onset of Grade 2+ and/or Grade 3+ Neurotoxicity as Assessed by NCI CTCAE Active Version
Description: Time to onset of grade 2+ neurotoxicity was defined as time from randomization to the first occurrence of grade 2+ neurotoxicity. Time to onset of grade 3+ neurotoxicity was defined as time from randomization to the first occurrence of grade 3+ neurotoxicity.
Time Frame: Up to 12 months from initiation of ixabepilone
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Overall
Number analyzed (Participants) | 0

4. Secondary Outcome: Proportion of Patients Undergoing Dose Reduction or Discontinuing Ixabepilone Secondary to Peripheral Neuropathy
Time Frame: Up to 12 months from initiation of ixabepilone
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Overall
Number analyzed (Participants) | 0

5. Secondary Outcome: Average Cumulative Ixabepilone Dose
Time Frame: Up to 12 months from initiation of ixabepilone
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Overall
Number analyzed (Participants) | 0

6. Secondary Outcome: Toxicity Profile of CaMg Per CTCAE Active Version
Time Frame: Up to 12 months from initiation of ixabepilone
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Overall
Number analyzed (Participants) | 0

7. Secondary Outcome: Incidence of the Acute Pain Syndrome (APS)
Description: APS was measured using the pain item which evaluated the aches/pains at its WORST in the last 24 hours in the scale of 0 to 10, with 0=no aches/pain and 10=aches/pains as bad as can be.
  The outcome measures for each subsequent cycle will be analyzed in a similar fashion.
Time Frame: Treatment initiation to day 21 (Cycle 1)
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Overall
Number analyzed (Participants) | 0

8. Secondary Outcome: Severity of the Acute Pain Syndrome (APS)
Description: as for outcome 7
Time Frame: Treatment initiation to day 21 (Cycle 1)
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Overall
Number analyzed (Participants) | 0

9. Secondary Outcome: Association Between the Ixabepilone-APS and Eventual Chemotherapy-induced Neuropathy
Description: Correlation coefficients will be produced relating the worst pain scores in the first cycle of therapy and the subsequent neuropathy scores as judged from the daily and weekly questions.
Time Frame: First cycle of therapy (up to 21 days)
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Overall
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Overall
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes